CLINICAL TRIAL: NCT01779167
Title: A Phase 2 Trial of Daily Alternating Thalidomide and Lenalidomide Plus Rituximab (ThRiL) for Patients With Previously Treated Waldenstrom Macroglobulinemia
Brief Title: Thalidomide, Lenalidomide, and Rituximab for Previously Treated Waldenstrom Macroglobulinemia
Acronym: THRiL for WM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1112012086; RV-WM-PI-0690 (Other Grant/Funding Number: Celegene)
Record Dates: First submitted 2013-01-07; First posted 2013-01-30 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Waldenstrom Macroglobulinemia
Keywords: WM
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Thalidomide; Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All Patients (Experimental): Daily alternating thalidomide and lenalidomide plus rituximab (ThRiL) in patients with previously treated WM
  Interventions: Drug: Thalidomide; Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Thalidomide — Thalidomide 50 mg (every ODD day of a 28 day cycle: Days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25 & 27)
Drug: Lenalidomide — Lenalidomide (every EVEN day of a 28 day cycle: Days 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26 & 28). Lenalidomide will be initiated at a starting dose of 5 mg.
  Other Names: Revlimid
Drug: Rituximab — Rituximab 375 mg/m2 IV on Days 1, 8, 15 and 22 (+/- 2 days) and then again on the same weekly x 4 schedule every 6th cycle thereafter (Cycle 7, 13, 19, etc).
  Other Names: Rituxan

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of daily alternating thalidomide and lenalidomide plus rituximab (ThRiL) in patients with previously treated Waldenstrom macroglobulunemia (WM). Thalidomide and lenalidomide are drugs that modulate the immune system and have been shown to bring about responses in subjects with WM. However, their use has been limited due to side effects. The investigators hypothesize that alternating doses of thalidomide and lenalidomide may alleviate the side effects while preserving the effectiveness of the therapies.

DETAILED DESCRIPTION:
Waldenstrom macroglobulinemia (WM) is an incurable B-cell lymphoproliferative disorder characterized by expansion of malignant B-lymphocytes and excessive production of monoclonal IgM. The survival and proliferation of the neoplastic WM cells is highly dependent on signals from the microenvironment. Thalidomide and lenalidomide are immunomodulatory agents with single agent activity in WM. Their use is limited by significant toxicities, including tumor flare (thalidomide and lenalidomide); sedation, constipation, and neuropathy (thalidomide); and cytopenias (lenalidomide). Alternating doses of thalidomide and lenalidomide may alleviate the toxicities, while preserving efficacy since the agents have non-overlapping toxicities and yet similar hypothesized mechanisms of action. Additionally, starting at a lower dose of lenalidomide than previously studied in WM may allow for improved tolerability. A pilot study of daily alternating therapy in subjects with chronic lymphocytic leukemia demonstrated that the two agents could be combined with non-overlapping toxicity. This phase II study aims to evaluate the efficacy and safety of daily alternating thalidomide and lenalidomide plus rituximab (ThRiL) in subjects with previously treated WM.

Subjects will receive thalidomide 50 mg every other day (i.e., every odd day: days 1, 3, 5, 7, 9, 11, 13, 15, 17, 19, 21, 23, 25 & 27 of a 28 day cycle) alternating with lenalidomide on every other day (i.e., every even day: days 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26 & 28 of a 28 day cycle), dosed based upon stepwise incremental dosing. Rituximab 375 mg/m2 will be administered on days 1, 8, 15 and 22 starting with Cycle 1 and then again on the same weekly x 4 schedule every 6th cycle thereafter (Cycles 7, 13, 19, etc).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of WM
* At least one prior systemic therapy
* Measurable disease, defined as quantifiable monoclonal IgM > 1000 mg/dL
* Active disease requiring therapy defined as at least one of the following five criteria:

  1. Rising IgM
  2. Hemoglobin < 20 g/dL
  3. Platelet count < 100 x 109/L
  4. Symptomatic or bulky lymphadenopathy or organomegaly
  5. Systemic manifestations of WM, including hyperviscosity, neuropathy, amyloidosis, cryoglobulinemia, B symptoms.
* note: subjects with symptomatic hyperviscosity or a serum viscosity of > 3.5 CP are eligible but should undergo plasmapheresis prior to initiation of treatment
* Understand and voluntarily sign an informed consent form
* Age >18 years at the time of signing the informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* ECOG performance status ≤ at study entry
* Laboratory test results within these ranges:

  1. Absolute neutrophil count ≥ 1000/mm³
  2. Platelet count ≥ 50,000/mm³
  3. Creatinine clearance of ≥ 30 mL/min by Cockroft-Gault formula.
  4. Total bilirubin ≤ 1.5 times the ULN, unless abnormality is the result of Gilbert's disease or the result of the WM
  5. AST (SGOT) and ALT (SGPT) ≤ 3 x ULN
* Disease free of prior malignancies for ≥ 2 years with exception of curatively treated basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
* All study participants must be registered into the mandatory RevAssist ® (RASP: RevAssist ® for Study Participants) and S.T.E.P.S. ® (P-TAP: Protocol Therapy Assistant Program) programs and be willing and able to comply with the requirements of RevAssist ® and S.T.E.P.S. ®.
* Females of childbearing potential (FCBP)† must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting treatment and again within 24 hours before the first dose of lenalidomide AND thalidomide. FCBP must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide and/or thalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All subjects must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure. See Appendix A: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.
* Able to take aspirin 81 or 325 mg daily or low molecular weight heparin as prophylactic anticoagulation, unless already on therapeutic anticoagulation. Subjects intolerant to ASA may use warfarin or low molecular weight heparin.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from providing informed consent.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Concurrent use of other anti-cancer agents or treatments
* Prior treatment with thalidomide or lenalidomide
* Active serious infection not controlled with antibiotics
* Autoimmune hemolytic anemia or thrombocytopenia requiring treatment
* Known positive for HIV
* Active infection with hepatitis B, defined by being positive for HepBsAg or Hep B DNA by PCR, or hepatitis C
* Pre-existing peripheral neuropathy > grade 2
* Pregnant or breast-feeding females. (Lactating females must agree not to breast feed while taking lenalidomide and/or thalidomide).
* Disease transformation to an aggressive histology
* Treatment for WM within the past 28 days
* Hypersensitivity to rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Martin, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Patients
Started | 4
Completed | 3
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 3
Age, Customized [Count of Participants; unit: Participants]
  50-59 | 1
  60-69 | 1
  80-89 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Demonstrate a Response (Complete, Partial, Minor) to Treatment
Description: Response criteria for subjects with WM is based upon the Consensus Panel Recommendations from the Third International Workshop on Waldenstrom Macroglobulinemia.
  Overall response rate (CR + PR + MR) measured at time of best response.
Time Frame: Approximately 24 months
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 3
participants | 0

2. Secondary Outcome: Number of Adverse Events Experienced With Alternating Thalidomide and Lenalidomide Plus Rituximab for Subjects With Previously Treated Waldenstrom's Macroglobulinemia
Description: Capture the number of adverse events experienced when combining thalidomide, lenalidomide, and rituximab in patients with previously treated WM
Time Frame: approximately 24 months per patient
Population: Data was not collected due to early termination.
Arm/Group | All Patients
Number analyzed (Participants) | 0

3. Secondary Outcome: Survival of Subjects Treated With THRiL for WM.
Description: Estimate overall survival of patients enrolled on THRiL for WM.
Time Frame: approximately 24 months per patient
Population: Data was not collected due to early termination.
Arm/Group | All Patients
Number analyzed (Participants) | 0

4. Secondary Outcome: Rate of Rituximab Related IgM Flare
Description: Estimate the rate of rituximab-related IgM flare
Time Frame: Approximately 24 months per patient
Population: Data was not collected due to early termination.
Arm/Group | All Patients
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Response
Description: Measure the time from initiating therapy to demonstrating response in WM.
Time Frame: approximately 24 months
Population: Data was not collected due to early termination.
Arm/Group | All Patients
Number analyzed (Participants) | 0

6. Secondary Outcome: Response Duration of Subjects Treated With THRiL for WM
Description: Measure response duration of patients enrolled on THRiL for WM
Time Frame: 24 months
Population: Data was not collected due to early termination.
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Patients (N=4)
Vasovagal Reaction (Nervous system disorders) | 1
Unconsciousness (General disorders) | 1
Gastrointestinal stromal tumor (Gastrointestinal disorders) | 1
Sick Sinus Syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Transient Ischemic Attacks (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=3)
Anemia (Blood and lymphatic system disorders) | 2 (5)
Neutropenia (Blood and lymphatic system disorders) | 3 (17)
Intermittent Creatinine increased (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3)
Hyperuricemia (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 2 (9)
Creatinine increased (Blood and lymphatic system disorders) | 2 (2)
Fatigue (worsened) (General disorders) | 1 (3)
aphasia (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes